CLINICAL TRIAL: NCT02666339
Title: Mélisses Garden: Effect of the Mediation by Care-garden on Anxious State in Adult Patients Hospitalized in Psychiatry (Prospective, Monocentric, Controlled, Randomized, Open in Two Parallel Groups Study)
Brief Title: Mélisses Garden: Effect on Anxious State in Adult Patients Hospitalized in Psychiatry
Acronym: JDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1508192; 2016-A00057-44 (Other: ANSM)
Record Dates: First submitted 2016-01-15; First posted 2016-01-28 (Estimated); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Psychiatric Decompensation
Keywords: Hortitherapy; Care-garden; Anxiety; Therapeutic alliance
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hortitherapy group (Experimental): Hortitherapy + Usual care
  Interventions: Behavioral: Hortitherapy
- Control group (Active Comparator): Usual care
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Usual care — Usual care : drug therapy, nurse and physician consultations.
  Arms: Control group
Behavioral: Hortitherapy — 2 hortitherapy sessions/week during 4 weeks, added at the usual care.
  Arms: Hortitherapy group

SUMMARY:
Each hospitalization leads to stress and anxiety. This is particularly true in psychiatry, because of "decompensation". That is why therapeutic treatments are delivered quickly to treat these symptoms and to allow a better relationship with patients. This relationship patients-nursing staff called "therapeutic alliance" is needed in psychiatry. Moreover, other treatments added to the therapeutic ones are used, like mediation, to increase the patients' state of health.

These last years, numerous studies were based on hortitherapy or care-gardens. It consists in the use of plants with a medical staff (for example nurses). A lot demonstrated the efficacy of the care-gardens, but most of them showed methodological weaknesses.

That is why the investigators would like to perform a randomized study, controlled, and they aim to demonstrate the efficacy of hortitherapy on anxiety in patients allowed in adult psychiatry for at least 4 weeks.

DETAILED DESCRIPTION:
Each hospitalization leads to stress and anxiety. This is particularly true in psychiatry, because of "decompensation" that increases anxiety and fear. That is why therapeutic treatments are delivered quickly to treat these symptoms and to allow a better relationship with patients. This relationship patients-nursing staff called "therapeutic alliance" is needed in psychiatry. Moreover, other treatments added to the therapeutic ones are used, like mediation, to increase the patients' state of health.

These last years, numerous studies were based on hortitherapy or care-gardens. It consists in the use of plants with a medical staff (for example nurses). A lot demonstrated the efficacy of the care-gardens, but most of them showed methodological weaknesses : no control group, no randomization, few patients. Furthermore, these studies were not performed with feared patients hospitalized in psychiatry.

That is why the investigators would like to perform a randomized study, controlled, and they aim to demonstrate the efficacy of hortitherapy on anxiety in patients allowed in adult psychiatry for at least 4 weeks. This study will be performed on 190 patients who will be included in one of these groups:

* Control group : only usual care
* Hortitherapy group : 2 hortitherapy sessions/week during 4 weeks, added at the usual care.

Anxiety will be evaluated with HAD-A scale that is a brief questionnaire (2 at 6 minutes). HAD-A is very sensitive at the modifications and allows to follow the evolution of the anxiety. This scale is easy to use by the nursing staff and shows an excellent reliability, by the way really adapted to this study. On another hand researchers will also focus on the effects on the therapeutic alliance and the persistence of the effects at week 8.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 18 years old
* Adult patient in complete hospitalization in psychiatry at CHU St-Etienne, with an anxiety score > 8 at HAD-A (cut off)
* Patient with hospitalization programmed for at least 1 month
* Patient able to start a mediation
* Antitetanic cover up to date (quick test performed before the randomization)
* Patients who have given their informed consent before participation in the study or for patients under supervision , informed consent of the guardian
* Patient affiliated or entitled to a social security scheme

Exclusion Criteria:

* Rejection of the randomization
* Inability to complete the scales whatever the cause of this failure (language other than French, mental retardation ...).
* Patient whose behavior evaluated by the psychiatrist does not allow the indication of a mediation.
* Patient who already participated in the mediation of horticultural therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
Effect of the mediation by care-garden on anxious state in adult patients hospitalized in psychiatry | 1 Month
  Score to HAD (anxiety scale)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine MASSOUBRE, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Joubert A, Jankowski-Cherrier B, Rossi A, Teyssier L, Suraud V, Presle E, Pommier R, Massoubre C, Verot E. Impact of horticultural therapy on patients admitted to psychiatric wards, a randomised, controlled and open trial. Sci Rep. 2024 Jun 22;14(1):14378. doi: 10.1038/s41598-024-65168-0. PMID 38909093